CLINICAL TRIAL: NCT04765605
Title: Guo's Subclavian Artery Reconstruction: The Prospective, Multiple Center Study of WeFlow-Tbranch Stent Graft System(GUEST Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hangzhou Endonom Medtech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WeFlow001
Record Dates: First submitted 2021-02-04; First posted 2021-02-21 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-08

CONDITIONS: Type B Aortic Dissection
Keywords: Type B Aortic Dissection; proximal left subclavian artery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WeFlow-Tbranch Stent Graft System (Experimental): Participants will be treated with WeFlow-Tbranch Stent Graft System
  Interventions: Device: WeFlow-Tbranch Stent Graft System

INTERVENTIONS:
Device: WeFlow-Tbranch Stent Graft System — The single-embedded branch thoracic aorta stent graft system consists of the thoracic aorta stent graft system and the branch stent system. The main chest embedded stent graft system consists of the main chest embedded stent graft and its system conveyor, and the branch stent system consists of branch stents and its conveyor. The main chest embedded stent graft and the branch stent are pre-installed in the conveyor

SUMMARY:
This study is a prospective, multiple center study to evaluate the safety and effectiveness of WeFlow-Tbranch single embedded branch thoracic aorta stent graft system manufactured by EndoNom Medtech (Hangzhou) Co., Ltd.

DETAILED DESCRIPTION:
This study is a prospective, multiple center study to evaluate the safety and effectiveness of WeFlow-Tbranch single embedded branch thoracic aorta stent graft system in the treatment of Stanford type B dissection of the proximal left subclavian artery. It is expected to complete the implantation of 120 patients in 29 centers within 12 months, and interim follow-up was conducted before discharge, 30 days after surgery, 6 months after surgery and 12 months after surgery, long-term follow-up will be performed at 24 months postoperatively, 36 months postoperatively, 48 months postoperatively and 60 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old, no gender limitation;
2. Able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the patient him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol;
3. Diagnosed as Stanford type B aortic dissection and needed reconstruction of the left subclavian artery;
4. The diameter of the proximal anchoring area (the aorta at the posterior edge of the left common carotid artery) range: 18～42mm;
5. The length of the proximal anchoring area (the distance from the rear edge of the left common carotid artery opening to the first breach) ≥15mm;
6. The distance between the left common carotid artery and the left subclavian artery ≥5mm;
7. The distance between the left vertebral artery and the opening of the left subclavian artery is ≥15mm, the diameter of the starting part of the left subclavian artery is 6～20mm
8. With proper femoral artery, iliac artery, and brachial artery access, endovascular treatment of the aorta can be performed.

Exclusion Criteria:

1. Pregnant, breastfeeding or cannot contraception during the trial period;
2. Participated in clinical trials of other drugs or devices during the same period;
3. The same operation requires intervention in other vascular diseases (such as coronary artery, renal artery, superior mesenteric artery, etc.), and the postoperative drug treatment plan is therefore affected;
4. Allergic to contrast agents, anesthetics, patches, and delivery materials;
5. Cannot tolerate anesthesia;
6. Severe liver, kidney, lung, and heart function abnormalities before surgery [Serum creatinine exceeds 2 times the upper limit of normal; Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeds 5 times the upper limit of normal; Serum total bilirubin (STB) more than 2 times the upper limit of normal; Left ventricular ejection fraction is lower than normal by cardiac color Doppler ultrasound examination];
7. True/false thoracic aortic aneurysm
8. History of myocardial infarction, TIA or cerebral infarction within the past 3 months;
9. Contraindications to antiplatelet drugs and anticoagulants
10. Life expectancy is less than 12 months (such as advanced malignant tumors)
11. Acute systemic infection
12. Severe stenosis or calcification in the anchoring area at the proximal end of the stent, easily lead to the stent graft difficult adherent
13. Investigator judged that not suitable for interventional treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Rate of no major adverse events within 30 days after surgery. | 30 days after operation
  Major adverse events within 30 days after operation refer to all-cause death, myocardial infarction, ischemic stroke, respiratory failure, liver failure, renal failure, intestinal necrosis, paraplegia, and amputation within 30 days after operation. Among them, renal failure refers to long-lasting dialysis, kidney transplantation, or other fatal results. Intestinal necrosis is intestinal ischemia that requires bowel resection or other fatal consequences. Severe lower limb ischemia refers to new severe limp or resting pain after surgery.
Treatment success rate of aortic dissection 12 months after operation | 12 months after operation
  The success rate of aortic dissection treatment at 12 months is a composite index, including immediate technical success after surgery and no displacement of the aorta and branch stent grafts in CTA 12 months after surgery, and no type I and type III endoleaks, the branch stent was unobstructed, and no second surgical intervention occurred during the follow-up period.

SECONDARY OUTCOMES:
All-cause mortality, aortic dissection-related mortality, serious adverse events, device-related adverse events, incidence of left upper limb ischemia. | 30 days, 6 months, and 12 months after operation
  1. All-cause mortality 30 days, 6 months, and 12 months after operation.
  2. Mortality related to aortic dissection 30 days, 6 months, and 12 months after operation.
  3. Incidence of serious adverse events 30 days, 6 months, and 12 months after operation.
  4. The incidence of device-related adverse events 30 days, 6 months, and 12 months after operation.
  5. Incidence of left upper limb ischemia 30 days, 6 months, and 12 months after operation.
The incidence of type I or type III endoleaks | during operation, 30 days after operation, 6 months, 12 months
  Record the endoleaks shown in the postoperative DSA or CTA images. Intraoperative endoleaks and adjuvant treatment are not recorded. Endoleaks that occurred after the completion of the operation and those that were not treated in the same subject at different follow-up stages were counted once.
Incidence of displacement of aorta and branch stent graft | 6 months and 12 months after surgery
  Observe and record CTA at 6 months and 12 months after operation to check the stent displacement, the main stent and branch stents are recorded and evaluated. Displacement was defined as the displacement of the node aorta and branch stent grafts by more than 10 mm compared to the 30th day after surgery.
Postoperative branch vessel patency rate | 30 days, 6 months, 12 months after surgery
  Observe and record CTA on the 30th day, 6 months, and 12 months after operation to evaluate the revascularization of branch vessels, whether there is occlusion, stenosis or thrombosis in the stent. Postoperative branch vessel stenosis ≤50% is considered unobstructed.
Success rate of remodeling of aortic dissection | 30 days, 6 months, 12 months after surgery
  Compare the results of CTA before operation and on the 30th day, 6th month and 12th month after operation, the expansion of the true lumen and the thrombosis of the false lumen at the coverage of the aortic dissection vascular stent to determine whether the blood vessel is successfully remodeled.
Incidence of conversion to thoracotomy or secondary interventional surgery due to aortic dissection | immediately after the surgery, 30 days after operation, 6 months, 12 months, 2~5 years
  To evaluate whether the subject was converted to thoracotomy or secondary interventional surgery due to aortic dissection.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Guo, Professor, Principal Investigator — Chinese PLA General Hospital
Locations (29):
- China (29):
  - Chinese PLA General Hospital, Beijing
  - Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing
  - Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Foshan First People's Hospital, Foshan
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Anhui Provincial Hospital, Hefei
  - Shandong Provincial Hospital, Jinan
  - The First People's Hospital of Yunnan Province, Kunming
  - Affiliated Hospital of Southwest Medical University, Luzhou
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Provincial People's Hospital, Nanjing
  - Nanjing Gulou Hospital, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Jiaotong University Affiliated Ninth People's Hospital, Shanghai
  - The Second Affiliated Hospital of Naval Medical University, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - The First Hospital of Hebei Medical University, Shijia Zhuang
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Bethune Hospital, Taiyuan
  - Tianjin Chest Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of PLA Air Force Military Medical University, Xi'an
  - Yantai Yuhuangding Hospital, Yantai
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No